CLINICAL TRIAL: NCT01835548
Title: A Randomized, Multicenter, Double-Blind, Placebo Controlled, Parallel Group Study of NT0102 in Children (Ages 6 12 Years) With Attention-Deficit Hyperactivity Disorder
Brief Title: NT0102 in the Treatment of Children With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neos Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NT0102.1004
Record Dates: First submitted 2013-04-08; First posted 2013-04-19 (Estimated); Results first posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2017-12

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NT0102 (Experimental): After the screening/washout period, all participants will receive study drug NT0102 once daily for 4 weeks during the dose optimization period. After completion of the dose optimization period, the optimized dose of the study drug will be selected, and participants will stay on that dose for 1 week (dose stabilization period). At the end of this period, participants will be randomized to a treatment. Participants in this arm will be given 20-60 mg of NT0102 as oral disintegrating tablet (ODT) once daily for one week during the double-blind treatment period.
  Interventions: Drug: NT0102
- Placebo (Placebo Comparator): After the screening/washout period, all participants will receive study drug NT0102 once daily for 4 weeks during the dose optimization period. After completion of the dose optimization period, the optimized dose of the study drug will be selected, and participants will stay on that dose for 1 week (dose stabilization period). At the end of this period, participants will be randomized to a treatment. Participants in this arm will be given placebo as matching ODT once daily for one week during the double-blind treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NT0102 — NT0102 (methylphenidate polistirex [MPP] extended release [XR] ODT) was given once daily at a dose equivalent to 20-60 mg methylphenidate hydrochloride.
  Arms: NT0102
Drug: Placebo — Matching ODT placebo was given once daily.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel group, Phase 3 trial to evaluate the safety and efficacy of NT0102 in the treatment of Attention Deficit Hyperactivity Disorder (ADHD) in pediatric patients 6 to 12 years of age in a laboratory classroom study.

ELIGIBILITY:
Inclusion Criteria:

* Currently being treated for ADHD

Exclusion Criteria:

* Other psychiatric diagnoses
* Significant cognitive impairment
* Chronic medical illnesses
* Structural cardiac defects
* Significant abnormal lab tests
* Taking disallowed medications
* Positive drug test

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Sikes, PhD, Study Director — Neos Tx
Locations (4):
- United States (4):
  - Florida Clinical Research Center, Bradenton, Florida
  - Florida Clinical Research Center, Maitland, Florida
  - Center for Psychiatry and Behavioral Medicine, Las Vegas, Nevada
  - Duke University, Durham, North Carolina

REFERENCES:
- [Derived] Childress AC, Kollins SH, Cutler AJ, Marraffino A, Sikes CR. Open-Label Dose Optimization of Methylphenidate Extended-Release Orally Disintegrating Tablet in a Laboratory Classroom Study of Children with Attention-Deficit/Hyperactivity Disorder. J Child Adolesc Psychopharmacol. 2021 Jun;31(5):342-349. doi: 10.1089/cap.2020.0142. Epub 2021 Jun 2. PMID 34081560
- [Derived] Childress AC, Kollins SH, Cutler AJ, Marraffino A, Sikes CR. Efficacy, Safety, and Tolerability of an Extended-Release Orally Disintegrating Methylphenidate Tablet in Children 6-12 Years of Age with Attention-Deficit/Hyperactivity Disorder in the Laboratory Classroom Setting. J Child Adolesc Psychopharmacol. 2017 Feb;27(1):66-74. doi: 10.1089/cap.2016.0002. Epub 2016 May 16. PMID 27183299

RESULTS

PARTICIPANT FLOW:
Groups:
- NT0102: After the screening/washout period, all participants received study drug NT0102 once daily for 4 weeks during the dose optimization period. After completion of the dose optimization period, the optimized dose of the study drug was selected, and participants were to stay on that dose for 1 week (dose stabilization period). At the end of this period, participants were randomized to a treatment. Participants in this arm were given 20-60 mg of NT0102 as oral disintegrating tablet (ODT) once daily for one week during the double-blind treatment period.
- Placebo: After the screening/washout period, all participants received study drug NT0102 once daily for 4 weeks during the dose optimization period. After completion of the dose optimization period, the optimized dose of the study drug was selected, and participants were to stay on that dose for 1 week (dose stabilization period). At the end of this period, participants were randomized to a treatment. Participants in this arm were given placebo as matching ODT once daily for one week during the double-blind treatment period.
- All Participants: All participants in the study went through the screening/washout period, then received study drug NT0102 once daily for 4 weeks during the dose optimization period. After completion of the dose optimization period, the optimized dose of the study drug was selected, and participants stayed on that dose for 1 week during the dose stabilization period before randomization into the double-blind treatment period.
Period: Screening/Washout Period
Arm/Group | NT0102 | Placebo | All Participants
Started | 0 | 0 | 87
Completed | 0 | 0 | 87
Not Completed | 0 | 0 | 0
Period: Dose Optimization Period
Arm/Group | NT0102 | Placebo | All Participants
Started | 0 | 0 | 87
Completed | 0 | 0 | 85
Not Completed | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Dose Stabilization Period
Arm/Group | NT0102 | Placebo | All Participants
Started | 0 | 0 | 85
Completed | 0 | 0 | 85
Not Completed | 0 | 0 | 0
Period: Double-Blind Treatment Period
Arm/Group | NT0102 | Placebo | All Participants
Started | 44 | 41 | 0
Completed | 44 | 39 | 0
Not Completed | 0 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) consisted of all participants randomized to treatment who had at least 1 post-dose Swanson, Kotkin, Agler, M-Flynn, and Pelham (SKAMP)-Combined treatment assessment during the classroom testing session on Visit 8. Participants were analyzed as randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | NT0102 | Placebo | Total
Number analyzed (Participants) | 43 | 39 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.1 (1.86) | 9.3 (1.64) | 9.2 (1.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 30 | 24 | 54

OUTCOME MEASURES:

1. Primary Outcome: Swanson, Kotkin, Agler, M-Flynn, and Pelham (SKAMP) Score
Description: The primary efficacy endpoint was derived from the SKAMP-Combined score calculated as the total score of all 13 items of the SKAMP-Combined score. The SKAMP-Combined score was obtained by summing up each item score where each item is rated on a 7-point impairment scale (0=normal to 6=maximal impairment) for a total possible score of 0 to 78. A lower score indicates less symptomatology (i.e., is better). The SKAMP was a rating scale that specifically measures the classroom manifestations of ADHD. The SKAMP ratings were completed for all subjects at baseline (pre-dose) and at 1, 3, 5, 7, 10, 12, and 13 hours post-dose on the classroom testing day (Visit 8). The primary analysis time point for the primary efficacy endpoint was the average of all post-dose SKAMP scores during the 13-hour period.
Time Frame: Visit 8 (Day 42)
Population: The full analysis set (FAS) consisted of all participants randomized to treatment who had at least 1 post-dose SKAMP-Combined treatment assessment during the classroom testing session on Visit 8. Participants were analyzed as randomized.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | NT0102
Number analyzed (Participants) | 39 | 43
score on a scale | 24.3 (9.47) | 17.3 (7.48)
Statistical Analysis 1: Comparison: Placebo vs NT0102; Test type: Superiority; p < 0.0001, ANCOVA; Least Square Mean Difference = -11.04, 95% CI 2-sided [-13.9 to -8.20], Standard Error of Mean 1.4239

2. Secondary Outcome: Onset of Effect
Description: Onset of effect was defined as the first time point at which NT0102 separates from placebo on SKAMP-Combined scores. A separation was defined as a statistically significant difference at the 5% level of active drug over placebo. Data was collected separately for NT0102 and Placebo arms and is reported as a comparison analysis of the two arms. This assessment was collected on the full classroom day, Visit 8.
Time Frame: Visit 8 (Day 42) at 1 hour (h), 3 h, 5 h, 7 h, 10 h, 12 h and 13 h
Population: FAS consisted of all participants randomized to treatment who had at least 1 post-dose SKAMP-Combined treatment assessment during the classroom testing session on Visit 8. Participants were analyzed as randomized.
Measure: Number; unit: hour
Groups:
- All Participants: Includes all participants from experimental and placebo comparator arms.
Arm/Group | All Participants
Number analyzed (Participants) | 82
hour | 1

3. Secondary Outcome: Duration of Effect
Description: Duration of effect was defined as the last time point at which NT0102 separates from placebo on SKAMP-Combined scores. A separation was defined as a statistically significant difference at the 5% level of active drug over placebo. Data was collected separately for NT0102 and Placebo arms, and is reported as a comparison analysis of the two arms. This assessment was collected on the full classroom day, Visit 8.
Time Frame: Visit 8 (Day 42) at 1 hour (h), 3 h, 5 h, 7 h, 10 h, 12 h and 13 h
Population: as for outcome 2
Measure: Number; unit: hour
Arm/Group | All Participants
Number analyzed (Participants) | 82
hour | 12

4. Secondary Outcome: The Average of the SKAMP-Attention Scores
Description: The SKAMP Rating Scale was comprised of 2 behavioral subscales, including the "Attention" subscale (4 items). The SKAMP-Attention subscore evaluates concentration in the classroom and is obtained by summing up each item score where each item is rated on a 7-point impairment scale (0=normal to 6=maximal impairment) for total possible combined score of 0 to 24. A lower score indicates less symptomatology (i.e. is better). The SKAMP-Attention subscores were derived from 20 minutes of direct observations of participant behavior. Ratings were based on the frequency and quality of behaviors.
Time Frame: Visit 8 (Day 42)
Population: The per-protocol set were a subset of the FAS consisting of those participants who satisfied all of the inclusion/exclusion criteria and who correctly received the treatment to which they were randomized.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- NT0102: After the screening/washout period, all participants received study drug NT0102 once daily for 4 weeks during the dose optimization period. After completion of the dose optimization period, the optimized dose of the study drug was selected, and participants were to stay on that dose for 1 week (dose stabilization period). At the end of this period, participants were randomized to a treatment. Participants in this arm were given 20-60 mg of NT0102 as ODT once daily for one week during the double-blind treatment period.
Arm/Group | Placebo | NT0102
Number analyzed (Participants) | 38 | 42
score on a scale | 12.2 (4.20) | 9.4 (3.42)

5. Secondary Outcome: The Average of the SKAMP-Deportment Scores
Description: The SKAMP Rating Scale is comprised of 2 behavioural subscales, including the "Deportment" subscale (4 items). The SKAMP-Deportment subscore evaluates behaviour in the classroom and is obtained by summing up each item score where each item is rated on a 7-point impairment scale (0=normal to 6=maximal impairment) for total possible combined score of 0 to 24. A lower score indicates less symptomatology (i.e. is better). The SKAMP-Attention subscores were derived from 20 minutes of direct observations of participant behaviour. Ratings were based on the frequency and quality of behaviours.
Time Frame: Visit 8 (Day 42)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | NT0102
Number analyzed (Participants) | 38 | 42
score on a scale | 12.5 (6.23) | 7.9 (5.26)

6. Secondary Outcome: The Average of the Permanent Product Measure of Performance - Attempted (PERMP-A) Score
Description: The PERMP consisted of 400 math problems and was graded as number of problems "Attempted" (PERMP-A) and number of problems "Correct." (PERMP-C). It was an objective measure of performance during the classroom testing day.
Time Frame: Visit 8 (Day 42)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of problems attempted
Arm/Group | Placebo | NT0102
Number analyzed (Participants) | 39 | 43
number of problems attempted | 82.0 (39.55) | 107.5 (57.53)

7. Secondary Outcome: The Average of the Permanent Product Measure of Performance - Correct (PERMP-C) Score
Description: as for outcome 6
Time Frame: Visit 8 (Day 42)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of problems correct
Arm/Group | Placebo | NT0102
Number analyzed (Participants) | 39 | 43
number of problems correct | 78.6 (40.60) | 104.1 (58.27)

8. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Visit 9 (Day 43)
Population: The safety population included all participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Optimization/Stabilization Phase: All participants received study drug NT0102 once daily for 4 weeks during the dose optimization period. After completion of the dose optimization period, the optimized dose of the study drug was selected, and participants were to stay on that dose for 1 week (dose stabilization period).
- Double-Blind Phase: Placebo: At the end of the stabilization period, participants were randomized to a treatment. Participants in this arm were given placebo as matching ODT once daily for one week during the double-blind treatment period.
- Double-Blind Phase: NT0102: At the end of the stabilization period, participants were randomized to a treatment. Participants in this arm were given 20-60 mg of NT0102 as ODT once daily for one week during the double-blind treatment period.
Arm/Group | Dose Optimization/Stabilization Phase | Double-Blind Phase: Placebo | Double-Blind Phase: NT0102
Number analyzed (Participants) | 87 | 41 | 44
Participants | 70 | 10 | 11

ADVERSE EVENTS:
Time Frame: Up to Visit 9 (Day 43)
Description: The safety population included all participants who took at least 1 dose of study drug. In the section "Other (Not Including Serious) Adverse Events" all events in the study are reported (frequency threshold 0%).
Arm/Group | Dose Optimization/Stabilization Phase | Double-Blind Phase: Placebo | Double-Blind Phase: NT0102
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/41 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/41 | 0/44
Other Adverse Events (participants affected / at risk) | 70/87 | 10/41 | 11/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Optimization/Stabilization Phase (N=87) | Double-Blind Phase: Placebo (N=41) | Double-Blind Phase: NT0102 (N=44)
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 2 | 0 | 0
Myopia (Eye disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 19 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0
Irritability (General disorders) | 6 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 10 | 3 | 4
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 2 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood pressure increased (Investigations) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 23 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 4 | 0 | 0
Headache (Nervous system disorders) | 17 | 1 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 3 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Affect lability (Psychiatric disorders) | 8 | 0 | 0
Emotional disorder (Psychiatric disorders) | 1 | 0 | 0
Initial insomnia (Psychiatric disorders) | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 11 | 0 | 0
Middle insomnia (Psychiatric disorders) | 1 | 0 | 0
Negativism (Psychiatric disorders) | 1 | 0 | 0
Tic (Psychiatric disorders) | 2 | 0 | 0
Trichotillomania (Psychiatric disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less